CLINICAL TRIAL: NCT05155085
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Subcutaneous Lirentelimab in Adult Subjects With Moderate-to-Severe Atopic Dermatitis Inadequately Controlled by Topical Treatments
Brief Title: A Study to Assess Subcutaneous Lirentelimab (AK002) in Atopic Dermatitis
Acronym: ATLAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer pursuing development
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK002-018
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis
Keywords: AD; Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema | interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lirentelimab (AK002) SC 300 mg (Experimental): Subjects in this arm will receive 7 doses of 300 mg of lirentelimab (AK002) administered subcutaneously every 2 weeks.
  Interventions: Drug: AK002
- Placebo (Other): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AK002 — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
  Other Names: Lirentelimab
  Arms: Lirentelimab (AK002) SC 300 mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of subcutaneous lirentelimab (AK002), given every 2 weeks for 7 doses, in adult subjects with moderate-to-severe AD inadequately controlled by topical treatments. Subjects who complete the randomized, double-blind, placebo-controlled treatment period may have the option to enroll in an open-label extension period and receive up to 7 doses of subcutaneous lirentelimab.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject is able to understand the information on the study, has the capacity to consent, and has provided written informed consent.
2. Male or female aged ≥18 and ≤80 years at the time of signing the informed consent form.
3. Chronic AD (as defined by the American Academy of Dermatology Consensus Criteria) (Eichenfield, 2014) that has been present for at least 3 years before the screening visit.
4. Documented recent history of inadequate response to treatment with topical medications such as topical corticosteroids, calcineurin inhibitors, JAK inhibitors, or PDE4 inhibitors (crisaborole) for at least 4 weeks in the 6 months prior to screening, or subjects for whom these topical treatments are otherwise medically inadvisable (e.g., because of side effects or safety risks).
5. Subjects who are biologic naive or biologic-exposed. Biologic-exposed includes patients who have demonstrated secondary loss of response, intolerance, or lack of continued access to biologics due to economic reasons.
6. EASI score of ≥16 at screening and at baseline.
7. Involvement of at least 10% or more of BSA at screening and at baseline.
8. An IGA score of 3 or above on a scale from 0-4 at screening and at baseline.
9. The subject should have applied a stable dose of non-medicated, non-prescription, topical emollient at least twice daily for 7 consecutive days immediately before the baseline visit.

Key Exclusion Criteria:

1. Current use of biologics for any indication.
2. Demonstrated lack of primary response to treatment with a biologic for the treatment of AD defined as no response to treatment despite complete adherence to the prescribed regimen for at least 3 months (primary non-responders).
3. Use of any of the following treatments within 4 weeks prior to the baseline visit or any condition that in the opinion of the Investigator is likely to require such treatment(s) during the first 4 weeks of study treatment: (i) phototherapy for AD; (ii) immunosuppressive or immunomodulatory drugs, including but not limited to systemic calcineurin inhibitors (e.g., cyclosporin, tacrolimus), mTOR inhibitors (e.g., sirolimus, everolimus), anti-metabolites (e.g., azathioprine, methotrexate, 6-mercaptopurine, leflunomide, mycophenolate mofetil), alkylating agents (e.g., cyclophosphamide), TNF inhibitors (e.g., infliximab, adalimumab), eosinophil depleting drugs (e.g., pramipexole), and systemic corticosteroids; (iii) oral JAK inhibitors within 8 weeks of the baseline visit.
4. Treatment with biologics: (i) any cell-depleting agents including but not limited to rituximab within 6 months prior to the baseline visit or until lymphocyte count returns to normal, whichever is longer; (ii) other biologics (e.g., dupilumab, omalizumab, etc) within 5 half-lives, if known, or 8 weeks prior to baseline visit, whichever is longer.
5. Use of any topical corticosteroids, topical calcineurin inhibitors, topical JAK inhibitors (e.g., ruxolitinib), or topical PDE4 inhibitors (crisaborole) for the treatment of AD within 1 week prior to the baseline visit.
6. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit.
7. Treatment with chemotherapy or radiotherapy in the preceding 6 months.
8. Presence of skin comorbidities/concomitant conditions that may interfere with study assessments or interpretation of study results.
9. Planned or anticipated use of any prohibited medications.
10. History of malignancy except carcinoma in situ in the cervix, early-stage prostate cancer, or non-melanoma skin cancers.
11. Any disease, condition (medical or surgical), or cardiac abnormality that in the opinion of the Investigator would place the subject at increased risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lee, MD, MPH, Study Director — Allakos Inc.
Locations (55):
- United States (40):
  - Allakos Investigational Site 218-034, Birmingham, Alabama
  - Allakos Investigational Site 218-074, Cullman, Alabama
  - Allakos Investigational Site 218-025, Gilbert, Arizona
  - Allakos Investigational Site 218-041, Scottsdale, Arizona
  - Allakos Investigational Site 218-072, Canoga Park, California
  - Allakos Investigational Site 218-056, Los Angeles, California
  - Allakos Investigational Site 218-073, San Diego, California
  - Allakos Investigational Site 218-051, San Francisco, California
  - Allakos Investigational Site 218-013, Santa Monica, California
  - Allakos Investigational Site 218-033, Santa Monica, California
  - Allakos Investigational Site 218-071, Colorado Springs, Colorado
  - Allakos Investigational Site 218-045, Washington D.C., District of Columbia
  - Allakos Investigational Site 218-018, Doral, Florida
  - Allakos Investigational Site 218-046, Greenacres City, Florida
  - Allakos Investigational Site 218-049, Jacksonville, Florida
  - Allakos Investigational Site 218-008, Miami, Florida
  - Allakos Investigational Site 218-048, Sarasota, Florida
  - Allakos Investigational Site 218-020, Tampa, Florida
  - Allakos Investigational Site 218-007, Tampa, Florida
  - Allakos Investigational Site 218-068, Lexington, Kentucky
  - Allakos Investigational Site 218-055, Crowley, Louisiana
  - Allakos Investigational Site 218-012, Towson, Maryland
  - Allakos Investigational Site 218-069, White Marsh, Maryland
  - Allakos Investigational Site 218-066, Boston, Massachusetts
  - Allakos Investigational Site 218-058, Dilworth, Minnesota
  - Allakos Investigational Site 218-063, Missoula, Montana
  - Allakos Investigational Site 218-032, Omaha, Nebraska
  - Allakos Investigational Site 218-026, Las Vegas, Nevada
  - Allakos Investigational Site 218-050, Las Vegas, Nevada
  - Allakos Investigational Site 218-029, Great Neck, New York
  - Allakos Investigational Site 218-053, Rochester, New York
  - Allakos Investigational Site 218-001, Cincinnati, Ohio
  - Allakos Investigational Site 218-062, Fairborn, Ohio
  - Allakos Investigational Site 218-003, Oklahoma City, Oklahoma
  - Allakos Investigational Site 218-015, Oklahoma City, Oklahoma
  - Allakos Investigational Site 218-061, Portland, Oregon
  - Allakos Investigational Site 218-010, Philadelphia, Pennsylvania
  - Allakos Investigational Site 218-052, Dallas, Texas
  - Allakos Investigational Site 218-047, Murray, Utah
  - Allakos Investigational Site 218-009, Seattle, Washington
- Germany (15):
  - Allakos Investigational Site 218-201, Berlin
  - Allakos Investigational Site 218-215, Darmstadt
  - Allakos Investigational Site 218-216, Darmstadt
  - Allakos Investigational Site 218-208, Dresden
  - Allakos Investigational Site 218-207, Erlangen
  - Allakos Investigational Site 218-212, Frankfurt am Main
  - Allakos Investigational Site 218-211, Gera
  - Allakos Investigational Site 218-203, Löhne
  - Allakos Investigational Site 218-210, Magdeburg
  - Allakos Investigational Site 218-204, Mainz
  - Allakos Investigational Site 218-213, Mainz
  - Allakos Investigational Site 218-218, Munich
  - Allakos Investigational Site 218-205, Osnabrück
  - Allakos Investigational Site 218-202, Recklinghausen
  - Allakos Investigational Site 218-209, Schwerin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 subjects who were enrolled in the main study received up to 7 doses of AK002 or placebo. 112 subjects from the main study continued into the open-label extension (OLE) period and received up to 7 doses of AK002.
Groups:
- AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE): For the main study period, subjects in this arm received up to 7 doses of 300 mg of lirentelimab (AK002) administered subcutaneously (SC) every 2 weeks.
  For the open-label extension (OLE) period, subjects who completed the main study and met eligibility criteria had the option to receive 7 doses of 300 mg AK002 SC.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
- Placebo (Main Study) - Placebo Rollover (OLE): For the main study period, subjects in this arm received up to 7 doses of placebo administered subcutaneously every 2 weeks.
  For the open-label extension (OLE) period, subjects who completed the main study and met the eligibility criteria had the option to rollover and receive 7 doses of 300 mg AK002 SC.
  Placebo: Placebo
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
Period: Main Study
Arm/Group | AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE) | Placebo (Main Study) - Placebo Rollover (OLE)
Started | 65 | 65
Completed | 57 | 58
Not Completed | 8 | 7
Period: Open-Label Extension
Arm/Group | AK002 SC 300 mg (Main Study) - AK002 Continuing (OLE) | Placebo (Main Study) - Placebo Rollover (OLE)
Started | 55 (2 subjects who completed the main study chose not to enter the open-label extension period.) | 57 (1 subject who completed the main study chose not to enter the open-label extension period.)
Completed | 32 | 36
Not Completed | 23 | 21

BASELINE CHARACTERISTICS:
Population: Baseline analysis is reported on the safety population of the main study period. Baseline information of OLE subjects is not reported since it is already captured as part of the main study population.
Groups:
- AK002 SC 300 mg (Main Study): Subjects in this arm received up to 7 doses of 300 mg of lirentelimab (AK002) administered subcutaneously every 2 weeks.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
- Placebo (Main Study): Subjects in this arm received up to 7 doses of placebo administered subcutaneously every 2 weeks.
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study) | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Median (Full Range); unit: years] | 41 [19 to 76] | 35 [19 to 75] | 38 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 20 | 44
  Not Hispanic or Latino | 38 | 42 | 80
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 23 | 38
  White | 43 | 35 | 78
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 53 | 106
  Germany | 12 | 12 | 24
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: Score on a scale] — The EASI score is a tool used to measure the extent (area) and severity of atopic dermatitis with respect to erythema, excoriation, induration, and lichenification over the 4 anatomic regions of the body: lower and upper extremities, trunk, and head. The total EASI score will be in a range from 0 to 72 points (from no disease to maximum disease severity).
  Score on a scale | 28.1 (7.5) | 30.1 (10.7) | 29.1 (9.2)
Investigator's Global Assessment (IGA) Score [Mean (Standard Deviation); unit: Score on a scale] — The Investigator's Global Assessment (IGA) is a 5-point scale that provides a global clinical assessment of AD severity ranging from 0 to 4 and assesses disease severity and clinical response using a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; and 4 = severe. The score is determined by ranking the extent of erythema and papulation/infiltration. A decrease in score relates to an improvement in signs and symptoms.
  Score on a scale | 3 (1) | 3 (1) | 3 (1)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieve 75% Improvement on the Eczema Area and Severity Index (EASI-75) at Week 14
Description: The EASI score is a tool used to measure the extent (area) and severity of atopic dermatitis with respect to erythema, excoriation, induration, and lichenification over the 4 anatomic regions of the body: lower and upper extremities, trunk, and head. The total EASI score will be in a range from 0 to 72 points (from no disease to maximum disease severity).
Time Frame: Baseline to Week 14
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Groups:
- AK002 SC 300 mg (Main Study): Subjects in this arm received up to 7 doses of 300 mg of lirentelimab (AK002) administered subcutaneously every 2 weeks in the main study.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
- Placebo (Main Study): Subjects in this arm received up to 7 doses of placebo administered subcutaneously every 2 weeks in the main study.
  Placebo: Placebo
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 61 | 61
percentage of participants | 23.0 | 18.0
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.4662, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.1, 95% CI 2-sided [-9.8 to 19.8]

2. Secondary Outcome: Percent Change in EASI From Baseline to Week 14
Description: as for outcome 1
Time Frame: Baseline to Week 14
Population: Modified Intent-to-Treat Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of change
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 61 | 61
Percentage of change | -36.0 (8.7) | -26.3 (8.7)
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.3968, Mixed Models Analysis; LSM Difference from Placebo = -9.7, 95% CI 2-sided [-32.2 to 12.9], Standard Error of Mean 11.4

3. Secondary Outcome: Proportion of Subjects Achieving an IGA Score of 0 or 1 and a 2-point Improvement at Week 14 vs Baseline
Description: The Investigator's Global Assessment (IGA) is a 5-point scale that provides a global clinical assessment of AD severity ranging from 0 to 4 and assesses disease severity and clinical response using a 5-point scale: 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; and 4 = severe. The score is determined by ranking the extent of erythema and papulation/infiltration. A decrease in score relates to an improvement in signs and symptoms.
Time Frame: Baseline to Week 14
Population: Modified Intent-to-Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study)
Number analyzed (Participants) | 61 | 61
percentage of participants | 11.5 | 8.2
Statistical Analysis 1: Comparison: AK002 SC 300 mg (Main Study) vs Placebo (Main Study); Test type: Superiority; p = 0.7625, Fisher Exact; Risk Difference (RD) = 3.3, 95% CI 2-sided [-15.2 to 21.6]

4. Other Pre Specified Outcome: Safety and Tolerability of up to 7 Doses of Open-label AK002 in Subjects With Atopic Dermatitis in the Open-label Extension Period
Description: Adverse events were assessed throughout the open-label extension period.
Time Frame: Through study completion, up to 38 weeks (open-label extension period)
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- AK002 Continuing (OLE): Subjects in this arm received AK002 in the main study and continued to receive up to 7 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
- Placebo Rollover (OLE): Subjects in this arm received placebo in the main study and rolled over to receive up to 7 doses of 300 mg AK002 SC in the open-label extension (OLE) period.
  Placebo: Placebo
  AK002: Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1(IgG1)monoclonal antibody directed against Siglec-8
Arm/Group | AK002 Continuing (OLE) | Placebo Rollover (OLE)
Number analyzed (Participants) | 55 | 57
Participants
  Subjects with ≥1 adverse events | 30 | 31
  Subjects with ≥1 treatment-related adverse events | 3 | 13
  Subjects with an adverse event leading to study drug discontinuation | 2 | 1
  Subjects with ≥1 serious adverse events | 2 | 0
  Subjects with ≥1 treatment-related serious adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, up to 38 weeks (open-label extension period)
Arm/Group | AK002 SC 300 mg (Main Study) | Placebo (Main Study) | AK002 Continuing (OLE) | Placebo Rollover (OLE)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/55 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/65 | 3/65 | 2/55 | 0/57
Other Adverse Events (participants affected / at risk) | 27/65 | 25/65 | 15/55 | 20/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 SC 300 mg (Main Study) (N=65) | Placebo (Main Study) (N=65) | AK002 Continuing (OLE) (N=55) | Placebo Rollover (OLE) (N=57)
Eczema herpeticum (Infections and infestations) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AK002 SC 300 mg (Main Study) (N=65) | Placebo (Main Study) (N=65) | AK002 Continuing (OLE) (N=55) | Placebo Rollover (OLE) (N=57)
Nasopharyngitis (Infections and infestations) | 3 | 4 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 2 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 12 | 4 | 0 | 9
Blood creatine phosphokinase increased (Investigations) | 0 | 5 | 1 | 1
Headache (Nervous system disorders) | 5 | 6 | 3 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 9 | 6 | 1
Injection site reaction (General disorders) | 1 | 1 | 0 | 6
Influenza (Infections and infestations) | 0 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Trial Agreement contains a limit on publication of results following completion of the trial. PIs are not allowed to publish results until a joint publication for the multicenter study or a set period of time. After that time, PIs may only publish results from their portion of the study.

DOCUMENTS (2):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT05155085/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT05155085/SAP_001.pdf